CLINICAL TRIAL: NCT02399969
Title: Battlefield Acupuncture for the Treatment of Low Back Pain in the Emergency Department
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCO 15-0360
Record Dates: First submitted 2015-03-23; First posted 2015-03-26 (Estimated); Last update posted 2016-05-05 (Estimated); Status verified 2016-05

CONDITIONS: Low Back Pain
Keywords: Low back pain; Acupuncture therapy; Acupuncture, ear
MeSH Terms: conditions — Low Back Pain | interventions — Acupuncture, Ear

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Battlefield Acupuncture Plus Standard of Care (Experimental): Patients with low back pain that will receive ear acupuncture based on the Battlefield Acupuncture protocol.
  Interventions: Other: Battlefield Acupuncture
- Standard of Care Alone (No Intervention): Patients with low back pain that will receive standard of care without study intervention.

INTERVENTIONS:
Other: Battlefield Acupuncture — Patients with low back pain will be randomized to receive Battlefield Acupuncture, ASP indwelling needles in 5 auricular (ear) points plus standard of care, or patients will be randomized to receive standard of care alone.
  Other Names: ear acupuncture, BFA
  Arms: Battlefield Acupuncture Plus Standard of Care

SUMMARY:
The purpose of this study is to study acupuncture for the treatment of low back pain in the emergency department. Current treatments for low back pain in the emergency department generally include pills or injections of medications to treat pain and relax muscles. However, it is known that many of these medications have risks and toxicities which may limit their safe use in some patients. Therefore, new types of treatments are needed.

Acupuncture is an ancient form of healing that has been practiced in some form for centuries. In modern times, acupuncture has been studied for the long-term treatment of low back pain and some research suggests it may be effective. However, very little research has examined the use of acupuncture for immediate pain relief in the emergency department.

This research will study a type of acupuncture called Battlefield Acupuncture (BFA). Battlefield acupuncture was designed by a physician in the US military with the purpose of providing immediate pain relief. It involves the placement of 5 small needles in each ear. The needles may be removed at any time. The hypothesis of this study is that battlefield acupuncture may improve mobility and pain of patients with low back pain in the emergency department.

DETAILED DESCRIPTION:
The researchers will review the chief complaints of patients arriving to the emergency department in epic. Subjects will be identified and recruited in the emergency department based on chief complaint of "back pain". Subjects will be approached by a researcher who will then recruit them to participate in the study using the attached informed consent form. Researchers will not be acting as treating physicians at the time of the study.

50 patients that present to the emergency setting with the complaint of low back pain will be randomized to standard care or standard care plus Battlefield Acupuncture. The patients randomized to receive Battlefield Acupuncture will receive the treatment according to the defined protocol, which involves placement of ASP indwelling needles in up to 5 auricular points. One ear will be selected, and the areas which will be needled will identified and prepped with alcohol to reduce risks of infection. Up to 5 sterile ASP semi- permanent needles will be placed. Treatments will be provided by MDs or PAs who have been trained to administer the Battlefield Acupuncture technique.

All patients will complete pre- and post- treatment surveys regarding their pain rating and functional limitation from pain. Additional data will be collected from EPIC regarding demographic information, medication administration, and length of stay.

Data will be collected from the subject at the time of enrollment, and again one hour following enrollment. No further data will be collected directly from subjects. Additional follow-up data regarding medications prescribed and length of stay will be collected from the chart after patient discharge.

ELIGIBILITY:
Inclusion criteria:

* adult
* English-speaking participants
* over the age of 18
* come to the emergency department with the chief complaint of low back pain.

Exclusion criteria:

* any focal neurological deficit
* prior back surgery, acute trauma,
* new weakness
* new loss bowel/bladder control
* back pain above T12
* receiving coumadin or plavix
* Pregnancy. Female patients will be offered pregnancy testing which they can elect to take.
* Temperature >38C,
* positive urinalysis (UTI or pregnancy). Urinalysis will not be requested if not deemed clinically relevant by the treating team, as this may delay patient care and discharge.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-03; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Get up and go test | baseline
  Time that a person takes to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down, will be monitored in seconds. If a person cannot get up in 30 seconds to ambulate, they will be cut off.
Get up and go test | immediately post-treatment in the BFA group only
  Time that a person takes to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down, will be monitored in seconds. If a person cannot get up in 30 seconds to ambulate, they will be cut off.
Get up and go test | 1 hour
  Time that a person takes to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down, will be monitored in seconds. If a person cannot get up in 30 seconds to ambulate, they will be cut off.

SECONDARY OUTCOMES:
Numeric Rating Scale (NRS) for Pain | baseline
  Patients will be asked "On a scale of 0 to 10, with 0 being no pain at all and 10 being the worst pain imaginable, how would you rate your pain right now"
Numeric Rating Scale (NRS) for Pain | immediately post-treatment in the BFA group only
  Patients will be asked "On a scale of 0 to 10, with 0 being no pain at all and 10 being the worst pain imaginable, how would you rate your pain right now"
Numeric Rating Scale (NRS) for Pain | 1 hour
  Patients will be asked "On a scale of 0 to 10, with 0 being no pain at all and 10 being the worst pain imaginable, how would you rate your pain right now"
Range of motion of the lumbar spine | baseline
  Active ROM (Flexion and Extension) will be measured using a goniometer
Range of motion of the lumbar spine | immediately post-treatment in the BFA group only
  Active ROM (Flexion and Extension) will be measured using a goniometer
Range of motion of the lumbar spine | 1 hour
  Active ROM (Flexion and Extension) will be measured using a goniometer

OTHER OUTCOMES:
Length of stay | up to 1 week
medications administered | up to 1 week
  Medications prescribed in the department and at discharge
Adverse events | up to 6 months
  Any adverse events reported by subjects will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Alex F Manini, MD, MS, FACMT, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Derived] Fox LM, Murakami M, Danesh H, Manini AF. Battlefield acupuncture to treat low back pain in the emergency department. Am J Emerg Med. 2018 Jun;36(6):1045-1048. doi: 10.1016/j.ajem.2018.02.038. Epub 2018 Feb 27. PMID 29550099